CLINICAL TRIAL: NCT06376019
Title: Evaluation of Occlusion and Disocclusion Time in Immediately Loaded Implant Supported Overdentures Supported by Two Splinted Versus Non Splinted Interforaminal Implants
Brief Title: Occlusion and Disocclusion Time in Immediately Loaded Overdentures Supported by Two Splinted Versus Non Splinted Interforaminal Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Mostafa Abdelfatah, associate professor of oral and maxillofacial prosthodontics, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDASU-RecID11352
Record Dates: First submitted 2024-04-17; First posted 2024-04-19 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Edentulous Jaw
MeSH Terms: conditions — Jaw, Edentulous | interventions — Denture, Complete

STUDY DESIGN:
Intervention Model Description: parallel assignment of the participants in ratio 1:1:1 will take place. For allocation concealment, opaque sealed envelopes will be used.
Masking Description: the statistician will be the only one to be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group CD (conventional complete denture group) (Placebo Comparator): patients will receive a conventional complete denture with no implant placement
  Interventions: Procedure: complete denture
- group IB (implant-supported overdenture with ball attachment) (Active Comparator): patients will receive an implant-supported overdenture with ball attachment. The overdenture will be relined by a soft liner.
  Interventions: Procedure: solitary Implant loading with ball attachment
- group II (implant-supported overdenture with an intraoral welded bar) (Active Comparator): patients will receive an implant-supported overdenture with an intraoral welded bar. The overdenture will be relined by a soft liner.
  Interventions: Procedure: splinted Implant loading with intra oral welding

INTERVENTIONS:
Procedure: solitary Implant loading with ball attachment — ball attachment will be attached to the dental implant on the day of implant placement
  Arms: group IB (implant-supported overdenture with ball attachment)
Procedure: splinted Implant loading with intra oral welding — Titanium bar will be welded to the dental implant on the day of implant placement
  Arms: group II (implant-supported overdenture with an intraoral welded bar)
Procedure: complete denture — Mucosa supported conventional complete denture will be fabricated without supporting implants
  Arms: group CD (conventional complete denture group)

SUMMARY:
complete denture wearers struggle to eat well with their dentures due to poor denture retention, stability, and occlusal disharmony. So, the current study protocol aims to compare the occlusion/ disocclusion time in immediately loaded implant retained overdentures supported by two interforaminal implants; splinted versus non splinted dental implants compared to the conventional complete denture.

DETAILED DESCRIPTION:
The gold standard treatment for completely edentulous patients is a removable complete denture, which satisfies patients functional and aesthetic requirements at a low cost. However, the main problem associated with a complete denture is the instability of the complete removable denture, especially the mandibular one. Implant-assisted overdentures over two or three implants are used as a treatment option to increase stability, function, and retention of the denture at a reasonable cost. The immediate loading protocol allows the placement of temporary restoration on the day of implant placement surgery. Pierluigi Mondani pioneered intraoral welding in the early 1970s as an approach to load patients immediately with resin prosthesis and weld titanium implants to a titanium bar in their mouths. The technique of intraoral welding provides rigid splinting in cases of immediate implant loading. Occlusal loads and stability of occlusion are important to consider in the immediate loading of implants to avoid implant biomechanical failures, marginal bone loss, or even complete loss of osseointegration. Quantitative analyzers like t-scans, which are pressure-sensitive films, and virtual technology give a precise method of assessing the sequence of time and occlusal contact force magnitude by converting qualitative data into quantitative parameters. So, the current study protocol aims to compare the occlusion/ disocclusion time in immediately loaded implant retained overdentures supported by two interforaminal implants; splinted versus non splinted dental implants compared to the conventional complete denture.

ELIGIBILITY:
Inclusion Criteria:

* completely edentulous patients
* non-smokers
* good oral hygiene
* motivated patients

Exclusion Criteria:

* major systemic diseases that may affect osseointegration as uncontrolled diabetes mellitus
* the need for extensive bone grafting in planned implant site
* pregnancy
* patients under bisphosphonate treatment
* limited mouth-opening for executing the implant surgery.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2024-04-25 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Assessment of occlusion/disocclusion time | 3 months
  occlusion/disocclusion time will be evaluated using a T scan device

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed MA Mohamed, BDS MSc MD, Principal Investigator — Ain Shams University
Locations (1):
- Faculty of Dentistry Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Raw statistical data will be available after publishing upon request from the corresponding author